CLINICAL TRIAL: NCT01206153
Title: Metformin for Treatment Antipsychotic Induced Amenorrhea in Female Schizophrenic Patients: a Double Blind, Placebo-controlled Study
Brief Title: Metformin for Treatment Antipsychotic Induced Amenorrhea in Female Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Jingping Zhao, the Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: RWu
Record Dates: First submitted 2010-09-13; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2008-02

CONDITIONS: Amenorrhea
MeSH Terms: conditions — Amenorrhea | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- metformin (Experimental)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin

SUMMARY:
Antipsychotics such as risperidone could induce amenorrhea in schizophrenic patients. The investigators conducted a randomized, placebo-controlled study to test the efficacy of metformin for antipsychotic induced amenorrhea in schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia patient
* amenorrhea for more than three months after antipsychotic treatment

Exclusion Criteria:

* liver or renal diseases
* pregnant or lactating women
* cardiovascular diseases
* hypertension or diabetes mellitus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
prolactin level
  the outcome measure assess a efficacy.

SECONDARY OUTCOMES:
fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Zhao, MD, Principal Investigator — Institute of Mental Health of The Second Xiangya Hospital, Central South University, 139# Renmin Middle Road，Changsha 410011, Hunan, P.R. China
Locations (1):
- Institute of Mental Health of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China